CLINICAL TRIAL: NCT02349074
Title: Digestive ENdoscopy afTeR Out-of-hospitAl Cardiac arresT
Acronym: ENTRACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Dr David GRIMALDI, Investigator coordinator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P13/30 ENTRACT; 2014-A00994-43 (Other: France : ANSM)
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Out-of-hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Digestive endoscopy (Experimental): Performed a systematic œsophago-gastro-duodenoscopy during Intensive Care Unit stay after out-of-hospital cardiac arrest
  Interventions: Procedure: Digestive endoscopy

INTERVENTIONS:
Procedure: Digestive endoscopy — Performed a systematic œsophago-gastro-duodenoscopy between 2 and 4 days after out-of-hospital cardiac arrest

SUMMARY:
Post-cardiac arrest ischemia/reperfusion phenomenon led to organs injury and failure. Among the different organs, gastro-intestinal tract injury could contribute to post-cardiac arrest shock.

The ischemic injury of the gastro-intestinal (GI) tractus is suggested by abnormalities in digestive biomarkers and by the frequent endotoxemia after CA. However, direct mucosal damage has not been clearly demonstrated after OHCA. The real incidence of ischemic lesions of GI tract and their potential involvement in the post-CA shock is therefore unknown.

We propose an original clinical research program aimed at rigorously determining the incidence of upper GI lesions after OHCA and analyzing their contribution to the severity of post-CA shock through a prospective, interventional, multicentric study

DETAILED DESCRIPTION:
The screening of the patients will be performed 2 to 4 days after their Intensive Care Unit (ICU) admission. Procedure and exams at the day of inclusion (day 0):

* collection of digestive symptoms
* carrying out the œsophago-gastro-duodenoscopy and establishment of a formal report with the eventual lesions and their ischemic nature.
* in the absence of contra-indication and upon final decision of the gastroscopist, systematic biopsies of fundic, antral and duodenal mucosa; contra-indication of biopsies are the presence of a vascular or haemorrhagic lesion and the coagulation disorders.
* Blood sample for H. pylori serology, and serum freezing. Urinary sample for urine freezing

Procedure and exams from day 1 to hospital discharge:

* Daily collection of digestive symptoms and needs for vasopressor support
* Sepsis-related Organ Failure Assessment (SOFA) score at day 2 & 5
* Cerebral Performance Category (CPC) score determination at hospital discharge In case of digestive symptoms after day 0 and in accordance with good clinical practice, a second gastroscopy and/or an abdominal Computed Tomography scan(CT-scan) and/or a colonoscopy will be performed at the physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient hospitalized for less than 5 days in a participating Intensive Unit Care following successfully resuscitated out-of-hospital cardiac arrest
* Patient still mechanically ventilated
* Hypothermia period over, corporal temperature > 36°C.
* Written consent from a next of kin

Exclusion Criteria:

* In-hospital cardiac arrest
* Patients extubated before gastroscopy
* Contra-indication of gastroscopy: suspicion of digestive perforation, severe bleeding diathesis despite coagulation products transfusion, or suspicion of Creutzfeldt-jacob disease
* Patients with cardiac valvular prosthesis or previous endocarditis
* Pregnancy, lactating women In case of severe coagulation disorders (platelet count < 30 G/L, International Normalized Ratio (INR) > 2) or heparin treatment or combined platelet inhibition treatment, the inclusion of the patient will be possible but digestive biopsies will not be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
To measure the incidence of upper digestive macroscopic lesions after out-of-hospital cardiac arrest | One day
  Performed a systematic œsophago-gastro-duodenoscopy between 2 and 4 days after the cardiac arrest

CONTACTS AND LOCATIONS:
Locations (9):
- Hospital Erasme, Brussels, Belgium
- France (8):
  - André Mignot Hospital, Intensive care unit, Le Chesnay, Les Yvelines
  - Cotentin Hospital, Medical intensive care unit, Cherbourg-Octeville
  - Hospital Louis Mourier, Colombes
  - Sud Francilien Hospital, Medicla care unit, Corbeil-Essonnes
  - Henri Mondor Hospital, Medical Intensive care unit, Créteil
  - Dupuytren hospital, Medical intensive care unit, Limoges
  - Orléans Hospital, Medical intensive care unit, Orléans
  - Cochin Hospital, Médical intensive care unit, Paris

REFERENCES:
- [Background] Dumas F, Grimaldi D, Zuber B, Fichet J, Charpentier J, Pene F, Vivien B, Varenne O, Carli P, Jouven X, Empana JP, Cariou A. Is hypothermia after cardiac arrest effective in both shockable and nonshockable patients?: insights from a large registry. Circulation. 2011 Mar 1;123(8):877-86. doi: 10.1161/CIRCULATIONAHA.110.987347. Epub 2011 Feb 14. PMID 21321156
- [Background] Dumas F, Cariou A, Manzo-Silberman S, Grimaldi D, Vivien B, Rosencher J, Empana JP, Carli P, Mira JP, Jouven X, Spaulding C. Immediate percutaneous coronary intervention is associated with better survival after out-of-hospital cardiac arrest: insights from the PROCAT (Parisian Region Out of hospital Cardiac ArresT) registry. Circ Cardiovasc Interv. 2010 Jun 1;3(3):200-7. doi: 10.1161/CIRCINTERVENTIONS.109.913665. Epub 2010 May 18. PMID 20484098
- [Background] Mongardon N, Dumas F, Ricome S, Grimaldi D, Hissem T, Pene F, Cariou A. Postcardiac arrest syndrome: from immediate resuscitation to long-term outcome. Ann Intensive Care. 2011 Nov 3;1(1):45. doi: 10.1186/2110-5820-1-45. PMID 22053891
- [Background] Lemiale V, Dumas F, Mongardon N, Giovanetti O, Charpentier J, Chiche JD, Carli P, Mira JP, Nolan J, Cariou A. Intensive care unit mortality after cardiac arrest: the relative contribution of shock and brain injury in a large cohort. Intensive Care Med. 2013 Nov;39(11):1972-80. doi: 10.1007/s00134-013-3043-4. Epub 2013 Aug 14. PMID 23942856
- [Background] Laver S, Farrow C, Turner D, Nolan J. Mode of death after admission to an intensive care unit following cardiac arrest. Intensive Care Med. 2004 Nov;30(11):2126-8. doi: 10.1007/s00134-004-2425-z. Epub 2004 Sep 9. PMID 15365608
- [Background] Laurent I, Monchi M, Chiche JD, Joly LM, Spaulding C, Bourgeois B, Cariou A, Rozenberg A, Carli P, Weber S, Dhainaut JF. Reversible myocardial dysfunction in survivors of out-of-hospital cardiac arrest. J Am Coll Cardiol. 2002 Dec 18;40(12):2110-6. doi: 10.1016/s0735-1097(02)02594-9. PMID 12505221
- [Background] Adrie C, Adib-Conquy M, Laurent I, Monchi M, Vinsonneau C, Fitting C, Fraisse F, Dinh-Xuan AT, Carli P, Spaulding C, Dhainaut JF, Cavaillon JM. Successful cardiopulmonary resuscitation after cardiac arrest as a "sepsis-like" syndrome. Circulation. 2002 Jul 30;106(5):562-8. doi: 10.1161/01.cir.0000023891.80661.ad. PMID 12147537
- [Background] Adrie C, Laurent I, Monchi M, Cariou A, Dhainaou JF, Spaulding C. Postresuscitation disease after cardiac arrest: a sepsis-like syndrome? Curr Opin Crit Care. 2004 Jun;10(3):208-12. doi: 10.1097/01.ccx.0000126090.06275.fe. PMID 15166838
- [Background] Hausenloy DJ, Yellon DM. Myocardial ischemia-reperfusion injury: a neglected therapeutic target. J Clin Invest. 2013 Jan;123(1):92-100. doi: 10.1172/JCI62874. Epub 2013 Jan 2. PMID 23281415
- [Background] Kawai T, Akira S. TLR signaling. Semin Immunol. 2007 Feb;19(1):24-32. doi: 10.1016/j.smim.2006.12.004. Epub 2007 Feb 1. PMID 17275323
- [Background] Suffredini AF, Fromm RE, Parker MM, Brenner M, Kovacs JA, Wesley RA, Parrillo JE. The cardiovascular response of normal humans to the administration of endotoxin. N Engl J Med. 1989 Aug 3;321(5):280-7. doi: 10.1056/NEJM198908033210503. PMID 2664516
- [Background] Balija TM, Lowry SF. Lipopolysaccharide and sepsis-associated myocardial dysfunction. Curr Opin Infect Dis. 2011 Jun;24(3):248-53. doi: 10.1097/QCO.0b013e32834536ce. PMID 21378563
- [Background] Zhou J, Huang WQ, Li C, Wu GY, Li YS, Wen SH, Lei WL, Liu KX. Intestinal ischemia/reperfusion enhances microglial activation and induces cerebral injury and memory dysfunction in rats. Crit Care Med. 2012 Aug;40(8):2438-48. doi: 10.1097/CCM.0b013e3182546855. PMID 22647410
- [Background] Marshall JC, Foster D, Vincent JL, Cook DJ, Cohen J, Dellinger RP, Opal S, Abraham E, Brett SJ, Smith T, Mehta S, Derzko A, Romaschin A; MEDIC study. Diagnostic and prognostic implications of endotoxemia in critical illness: results of the MEDIC study. J Infect Dis. 2004 Aug 1;190(3):527-34. doi: 10.1086/422254. Epub 2004 Jul 2. PMID 15243928
- [Background] Korth U, Krieter H, Denz C, Janke C, Ellinger K, Bertsch T, Henn C, Klein J. Intestinal ischaemia during cardiac arrest and resuscitation: comparative analysis of extracellular metabolites by microdialysis. Resuscitation. 2003 Aug;58(2):209-17. doi: 10.1016/s0300-9572(03)00119-9. PMID 12909384
- [Background] Gill RS, Lee TF, Sergi C, Bigam DL, Cheung PY. Early versus delayed cyclosporine treatment in cardiac recovery and intestinal injury during resuscitation of asphyxiated newborn piglets. Intensive Care Med. 2012 Jul;38(7):1215-23. doi: 10.1007/s00134-012-2577-1. Epub 2012 May 10. PMID 22572838
- [Background] Albrecht M, Gruenewald M, Zitta K, Zacharowski K, Scholz J, Bein B, Meybohm P. Hypothermia and anesthetic postconditioning influence the expression and activity of small intestinal proteins possibly involved in ischemia/reperfusion-mediated events following cardiopulmonary resuscitation. Resuscitation. 2012 Jan;83(1):113-8. doi: 10.1016/j.resuscitation.2011.06.038. Epub 2011 Jul 18. PMID 21763251
- [Background] Gill RS, Manouchehri N, Lee TF, Cho WJ, Thiesen A, Churchill T, Bigam DL, Cheung PY. Cyclosporine treatment improves mesenteric perfusion and attenuates necrotizing enterocolitis (NEC)-like intestinal injury in asphyxiated newborn piglets during reoxygenation. Intensive Care Med. 2012 Mar;38(3):482-90. doi: 10.1007/s00134-011-2436-5. Epub 2011 Dec 6. PMID 22143394
- [Background] Bedell SE, Fulton EJ. Unexpected findings and complications at autopsy after cardiopulmonary resuscitation (CPR). Arch Intern Med. 1986 Sep;146(9):1725-8. PMID 3753112
- [Background] Piton G, Barbot O, Manzon C, Moronval F, Patry C, Navellou JC, Belle E, Capellier G. Acute ischemic pancreatitis following cardiac arrest: a case report. JOP. 2010 Sep 6;11(5):456-9. PMID 20818115
- [Background] Gaussorgues P, Gueugniaud PY, Vedrinne JM, Salord F, Mercatello A, Robert D. Bacteremia following cardiac arrest and cardiopulmonary resuscitation. Intensive Care Med. 1988;14(5):575-7. doi: 10.1007/BF00263532. PMID 3221011
- [Background] Grootjans J, Lenaerts K, Derikx JP, Matthijsen RA, de Bruine AP, van Bijnen AA, van Dam RM, Dejong CH, Buurman WA. Human intestinal ischemia-reperfusion-induced inflammation characterized: experiences from a new translational model. Am J Pathol. 2010 May;176(5):2283-91. doi: 10.2353/ajpath.2010.091069. Epub 2010 Mar 26. PMID 20348235
- [Background] Thuijls G, van Wijck K, Grootjans J, Derikx JP, van Bijnen AA, Heineman E, Dejong CH, Buurman WA, Poeze M. Early diagnosis of intestinal ischemia using urinary and plasma fatty acid binding proteins. Ann Surg. 2011 Feb;253(2):303-8. doi: 10.1097/SLA.0b013e318207a767. PMID 21245670
- [Background] Crenn P, Messing B, Cynober L. Citrulline as a biomarker of intestinal failure due to enterocyte mass reduction. Clin Nutr. 2008 Jun;27(3):328-39. doi: 10.1016/j.clnu.2008.02.005. Epub 2008 Apr 28. PMID 18440672
- [Background] Grimaldi D, Guivarch E, Neveux N, Fichet J, Pene F, Marx JS, Chiche JD, Cynober L, Mira JP, Cariou A. Markers of intestinal injury are associated with endotoxemia in successfully resuscitated patients. Resuscitation. 2013 Jan;84(1):60-5. doi: 10.1016/j.resuscitation.2012.06.010. Epub 2012 Jun 26. PMID 22743354
- [Background] L'Her E, Cassaz C, Le Gal G, Cholet F, Renault A, Boles JM. Gut dysfunction and endoscopic lesions after out-of-hospital cardiac arrest. Resuscitation. 2005 Sep;66(3):331-4. doi: 10.1016/j.resuscitation.2005.03.016. PMID 16039032
- [Background] Jacobs I, Nadkarni V, Bahr J, Berg RA, Billi JE, Bossaert L, Cassan P, Coovadia A, D'Este K, Finn J, Halperin H, Handley A, Herlitz J, Hickey R, Idris A, Kloeck W, Larkin GL, Mancini ME, Mason P, Mears G, Monsieurs K, Montgomery W, Morley P, Nichol G, Nolan J, Okada K, Perlman J, Shuster M, Steen PA, Sterz F, Tibballs J, Timerman S, Truitt T, Zideman D; International Liason Committee on Resusitation. Cardiac arrest and cardiopulmonary resuscitation outcome reports: update and simplification of the Utstein templates for resuscitation registries. A statement for healthcare professionals from a task force of the international liaison committee on resuscitation (American Heart Association, European Resuscitation Council, Australian Resuscitation Council, New Zealand Resuscitation Council, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Southern Africa). Resuscitation. 2004 Dec;63(3):233-49. doi: 10.1016/j.resuscitation.2004.09.008. PMID 15582757
- [Background] Savoye G, Ben Soussan E, Hochain P, Lerebours E. [How and how far to investigate ischemic colitis?]. Gastroenterol Clin Biol. 2002 May;26(5 Suppl):B12-23. No abstract available. French. PMID 12068266
- [Derived] Grimaldi D, Legriel S, Pichon N, Colardelle P, Leblanc S, Canoui-Poitrine F, Ben Hadj Salem O, Muller G, de Prost N, Herrmann S, Marque S, Baron A, Sauneuf B, Messika J, Dior M, Creteur J, Bedos JP, Boutin E, Cariou A. Ischemic injury of the upper gastrointestinal tract after out-of-hospital cardiac arrest: a prospective, multicenter study. Crit Care. 2022 Mar 14;26(1):59. doi: 10.1186/s13054-022-03939-9. PMID 35287719